CLINICAL TRIAL: NCT06848062
Title: Validation of the Paris (Functional Coccydynia Effect) Pain Questionnaire for Coccydynia: A Study on Reliability and Validity in the Turkish Population
Brief Title: Validation of the Paris (Functional Coccydynia Effect) Pain Questionnaire
Acronym: Coccydynia
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aslinur Keles Ercisli, MD, Principal investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: 2024/12-12/39
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Coccydynia; Coccyx Disorder; Coccyx Injury
Keywords: coccyx; coccydynia; Paris Pain Questionnaire; validation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to validate and assess the reliability of the Turkish version of the Paris Pain Questionnaire (PPQ) in patients with coccydynia. The PPQ was developed by Dr. Jean-Yves Maigne as a condition-specific tool to evaluate pain severity and functional limitations in individuals with coccydynia. This study follows a cross-sectional observational design and includes 105 participants. The psychometric properties of the Turkish version will be assessed through internal consistency (Cronbach's alpha), test-retest reliability (intraclass correlation coefficient - ICC), and construct validity. The results will determine whether the PPQ is a valid and reliable tool for use in Turkish-speaking populations with coccydynia.

DETAILED DESCRIPTION:
Coccydynia refers to pain localized in the coccyx and surrounding areas without radiation, significantly affecting quality of life. The condition was first described in 1588, and in 1950, Schapiro referred to it as "television disease." Rectal palpation revealing tenderness in the coccyx strongly supports the diagnosis of coccydynia. Symptoms typically worsen while sitting (especially on hard surfaces), transitioning from sitting to standing, and prolonged standing. Although its etiology remains uncertain, the most common risk factors include internal and external trauma, such as falls and childbirth. While idiopathic cases may also occur, the risk of developing coccydynia is higher in women and individuals with obesity. Coccyx morphology and hypermobility are closely associated with coccydynia, and degenerative changes in the intercoccygeal discs have been implicated as a cause in 41% of idiopathic cases and 44% of traumatic cases. Tumors such as chordoma, osteoid osteoma, and notochordal cell tumors, as well as infections, are other potential causes.

Anteroposterior (AP) and lateral radiographs are the primary imaging modalities used to rule out these conditions and investigate predisposing factors for coccydynia, such as bone spicules, retroverted coccyx, coccygeal subluxation, or scoliosis. Radiographs are also valuable for identifying fractures or dislocations resulting from trauma. Additionally, angular mobility evaluations are performed using dynamic imaging techniques.

Clinical decision-making relies on valid and reliable outcome measures. These measures assess disability levels, functional impairment, treatment effectiveness, and disease progression over time. To be clinically meaningful, an outcome measure must be easy to complete and score, valid, reliable, and responsive to changes. The Oswestry Disability Index (ODI) is a valid, reliable, and responsive assessment tool specifically designed for low back pain. Although it has been widely used in studies assessing disability in coccydynia, it does not include coccydynia-specific functional limitations, such as "pain while transitioning from sitting to standing." Furthermore, ODI includes questions that assess leg pain, which is not relevant to coccydynia.

Similarly, quality of life is commonly assessed using the Short Form-12 (SF-12) in coccydynia research. However, SF-12 is a general health-related quality-of-life measure, rather than a condition-specific tool. Additionally, the Numeric Rating Scale (NRS) has long been used for pain assessment, and despite some criticisms, its use alongside additional questions provides valuable insights.

Assessing coccydynia requires the evaluation of pain and its functional impact, along with condition-specific disability questionnaires. The Paris Pain Questionnaire (Functional Impact of Coccydynia Pain Questionnaire) was developed by Jean-Yves Maigne in 2006 as a condition-specific tool. However, its reliability and validity have not been formally established.[6] While it has not been widely used in subsequent studies, it was reintroduced in 2021 by Jean-Yves Maigne and his team in another study on coccydynia assessment. In this study, a modification was made to the original questionnaire by incorporating pain onset during sitting. Unlike other questionnaires, the Paris Pain Questionnaire assesses aspects of pain that impact daily life, including pain while sitting (beyond intensity alone, as measured by NRS), transitioning from sitting to standing (highly specific to coccydynia with radiological findings), walking, nighttime pain (which is common in severe coccydynia), and pain during travel (a key indicator of coccygeal pain sensitivity). However, a formal validation and reliability study for this questionnaire has not been conducted to date.

This study aims to:

Translate the Paris Pain Questionnaire (Functional Impact of Coccydynia Pain Questionnaire) from English to Turkish.

Assess its validity and test-retest reliability (intra-rater reliability) in the Turkish-speaking population.

The Paris Pain Questionnaire was developed by Jean-Yves Maigne and his team and has been used in their clinical research; however, a formal reliability study has never been conducted. Currently, there is no standardized assessment tool specifically designed for coccydynia, and most studies rely on general low back pain measures.

Validating the Paris Pain Questionnaire is crucial for future research on coccydynia, as it provides a condition-specific measure of functional impact and pain severity. This study represents the first attempt to validate and establish the reliability of the Paris Pain Questionnaire, making it a valuable tool for clinicians and researchers. The Turkish validity and reliability study of this questionnaire will allow healthcare providers to use this unique assessment tool in Turkish-speaking patients with coccydynia.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years
* Diagnosis of coccydynia confirmed through clinical and radiological evaluation
* Ability to read and understand Turkish
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Presence of other conditions causing pelvic or rectal pain (e.g., endometriosis, ectopic pregnancy, hemorrhoids, rectal carcinoma)
* Severe psychiatric disorders (e.g., psychosis, major depression within the last 30 days)
* Neurological disorders affecting the pelvic region or lower back
* History of surgery or trauma to the coccygeal area within the past 90 days
* Primary complaints of low back pain rather than coccydynia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with coccydynia
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Internal Consistency (Cronbach's Alpha) | Baseline
  Internal consistency of the Turkish PPQ will be assessed using Cronbach's alpha.
Test-Retest Reliability (ICC) | Baseline and 3-day follow-up
  Intraclass correlation coefficient (ICC) will be calculated to assess reliability over time.

SECONDARY OUTCOMES:
Construct Validity (Pearson Correlation) | Baseline
  PPQ scores will be correlated with the Oswestry Disability Index (ODI), Numeric Rating Scale (NRS), and Short Form-12 (SF-12).
Factor Analysis | Baseline
  Exploratory factor analysis will be conducted to evaluate the structural validity of the Turkish PPQ

CONTACTS AND LOCATIONS:
Overall Officials: Aslinur Keles Ercisli, M. D., Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided